CLINICAL TRIAL: NCT05271045
Title: Formulation of Canola Oil With Vitamins A and D and γ-oryzanol and Evaluation of the Efficacy of Its Consumption Compared to Canola and Sunflower Oil Without γoryzanol in Adults With Type 2 Diabetes: a Randomized Controlled Clinical Trial
Brief Title: Assessment of the Efficacy of Vitamins A and D and γ-oryzanol-fortified Canola Oil in Adults With Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Tirang R. Neyestani, Ph.D., Prof., National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 25
Record Dates: First submitted 2022-02-27; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Diabetes
Keywords: vitamin A; vitamin D; γ-oryzanol; fortified oil
MeSH Terms: conditions — Diabetes Mellitus | interventions — Fumigant 93

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- fortified canola oil with vitamins A and D and γ-oryzanol (Experimental): daily intake of fortified canola oil (385 IU vitamin D/ 30g & 154 IU vitamin A/30 g & 2130 ppm γ-oryzanol/30g)
  Interventions: Dietary Supplement: fortified canola oil with vitamins A and D and γ-oryzanol
- fortified canola oil with vitamins A and D (Active Comparator): daily intake of fortified canola oil (385 IU vitamin D/ 30g & 154 IU vitamin A/30 g)
  Interventions: Dietary Supplement: Active comparator
- fortified sunflower oil with vitamins A and D (Placebo Comparator): daily intake of fortified sunflower oil (385 IU vitamin D/ 30g & 154 IU vitamin A/30 g)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: fortified canola oil with vitamins A and D and γ-oryzanol — 30 g fortified canola oil with vitamins A and D and γ-oryzanol
  Arms: fortified canola oil with vitamins A and D and γ-oryzanol
Dietary Supplement: Active comparator — 30 g fortified canola oil with vitamins A and D
  Arms: fortified canola oil with vitamins A and D
Dietary Supplement: Placebo — 30 g fortified sunflower oil with vitamins A and D
  Arms: fortified sunflower oil with vitamins A and D

SUMMARY:
The aim of this study is to evaluate the efficacy of daily intake of fortified canola oil with vitamins A and D and γ-oryzanol on anthropometric, inflammatory, immunity, appetite and metabolic indicators of adults with type 2 diabetes compared to canola and sunflower oil without γoryzanol.

DETAILED DESCRIPTION:
Ninety confirmed type 2 diabetes patients aged 20-65 years old will be selected. Participants who change their usual medicine intake or make any changes in their diet and lifestyle that could alter the effectiveness of the intervention as well as those who do not use the fortified oil for three consecutive days or do not use the fortified oil for more than ten days throughout the intervention will be excluded. Subjects will be assigned randomly to one of the three intervention groups: 1.fortified canola oil with vitamins A and D and γ-oryzanol , 2. fortified canola oil with vitamins A and D, 3. fortified sunflower oil with vitamins A and D. Each participant will consume 30 g of oil every day for 2 months.

At the first and last visits, dietary and laboratory assessments will be performed for all subjects. The primary outcomes are the improvement of anthropometric, inflammatory, immunity, appetite, glycemic, and lipidemic markers of adults with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetic patients with fasting blood sugar above 100 mg/dL or hemoglobin A1c above 6% in the last test
2. Age between 20 to 65 years
3. No use of insulin

Exclusion Criteria:

1. Changing usual medicine intake or making any changes in diet and lifestyle that could alter the effectiveness of the intervention
2. Not using the fortified oil for three consecutive days or not using the fortified oil for more than ten days throughout the intervention period

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
serum glucose (mg/dL) | 8 weeks
  Fasting serum glucose level
serum HbA1c (mg/dL) | 8 weeks
  Fasting serum HbA1c level

SECONDARY OUTCOMES:
Weight (Kg) | 8 weeks
  Subject's weight wearing light clothing
Body Mass Index (Kg/m2) | 8 weeks
  weight (kg) divided by the square of height (m)
Waist circumference (cm) | 8 weeks
  the measurement at the midpoint between the lowest rib and the iliac crest
25-hydroxyvitamin D (nmol/L) | 8 weeks
  Fasting serum 25-hydroxyvitamin D level
serum triglyceride (mg/dL) | 8 weeks
  Fasting serum triglyceride level
serum total cholesterol (mg/dL) | 8 weeks
  Fasting serum total cholesterol level
serum LDL (mg/dL) | 8 weeks
  Fasting serum low density lipoprotein level
serum HDL (mg/dL) | 8 weeks
  Fasting serum high density lipoprotein level
serum insulin (pg/mL) | 8 weeks
  Fasting serum insulin level
serum BUN (mg/dL) | 8 weeks
  Fasting serum BUN level
serum creatinine (mg/dL) | 8 weeks
  Fasting serum creatinine level
serum leptin (pg/mL) | 8 weeks
  Fasting serum leptin level
serum grelin (pg/mL) | 8 weeks
  Fasting serum grelin level
serum hsCRP (pg/mL) | 8 weeks
  Fasting serum high sensitivity c-reactive protein level
serum IL-6 (pg/mL) | 8 weeks
  Fasting serum Interleukin-6 level
serum IL-1β (pg/mL) | 8 weeks
  Fasting serum Interleukin-1β level
serum INF-γ (pg/mL) | 8 weeks
  Fasting serum INF-γ level
salivary sIg-A (pg/mL) | 8 weeks
  Fasting Salivary Secretory Immunoglobulin A
ox-LDL (mg/dL) | 8 weeks
  Fasting oxidized low density lipoprotein level
MDA (mg/dL) | 8 weeks
  Fasting serum malondialdehyde level
TAC (mg/dL) | 8 weeks
  Fasting serum total antioxidant capacity level

CONTACTS AND LOCATIONS:
Overall Officials: Tirang R. Neyestani, PhD, Study Chair — NationalNFTI, SBMU, Tehran, Iran
Locations (1):
- Laboratory of Nutrition Research, National Nutrition and Food Technology Research Institute (NNFTRI) and Faculty of Nutrition Science and Food Technology, Shahid Beheshti University of Medical Sciences, Tehran, Iran, Tehran, Iran

REFERENCES:
- [Derived] Nikooyeh B, Zargaraan A, Ebrahimof S, Kalayi A, Zahedirad M, Yazdani H, Rismanchi M, Karami T, Khazraei M, Jafarpour A, Neyestani TR. Added gamma-oryzanol boosted anti-inflammatory effects of canola oil in adult subjects with type 2 diabetes: a randomized controlled clinical trial. Eur J Nutr. 2024 Mar;63(2):425-433. doi: 10.1007/s00394-023-03275-w. Epub 2023 Nov 16. PMID 37971692
- [Derived] Nikooyeh B, Zargaraan A, Ebrahimof S, Kalayi A, Zahedirad M, Yazdani H, Rismanchi M, Karami T, Khazraei M, Jafarpour A, Neyestani TR. Daily consumption of gamma-oryzanol-fortified canola oil, compared with unfortified canola and sunflower oils, resulted in a better improvement of certain cardiometabolic biomarkers of adult subjects with type 2 diabetes: a randomized controlled clinical trial. Eur J Med Res. 2023 Oct 10;28(1):416. doi: 10.1186/s40001-023-01409-8. PMID 37817285